CLINICAL TRIAL: NCT06062082
Title: What is Intraoperative Hemodynamic Instability During Unilateral Adrenalectomy for Pheochromocytoma: an Observational Study
Brief Title: Intraoperative Hemodynamic Instability During Unilateral Adrenalectomy for Pheochromocytoma
Acronym: HEMODADRE
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Laurent BRUNAUD, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: reference 2020PI123
Record Dates: First submitted 2022-07-06; First posted 2023-10-02 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Pheochromocytoma; Non-Secretory Adrenal Adenoma
Keywords: adrenalectomy
MeSH Terms: conditions — Pheochromocytoma | interventions — Adrenalectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pheochromocytoma: Patients operated on for pheochromocytoma by unilateral adrenalectomy
  Interventions: Procedure: adrenalectomy
- Control: Patients operated on for adrenal tumor other than pheochromocytoma by unilateral adrenalectomy
  Interventions: Procedure: adrenalectomy

INTERVENTIONS:
Procedure: adrenalectomy — laparoscopic exeresis of the adrenal gland

SUMMARY:
Pheochromocytomas are tumors of the adrenal gland that develop from cells producing adrenaline and noradrenaline. Consequently, intraoperative blood pressure variations (hypertensive and hypotensive episodes) are characteristic of pheochromocytoma surgery, when these tumors are removed. However, recommendations for the management of these tumors are based on data essentially dating from the 1960s-1990s. Since then, anesthesia and surgery for patients with pheochromocytoma have evolved considerably, and have become more effective with time. In these circumstances, a review of the current situation is necessary. The aim of this study is to investigate the intraoperative hemodynamic changes observed in patients undergoing adrenalectomy for pheochromocytoma, comparing them with the hemodynamic profile observed in patients undergoing adrenal surgery for a pathology other than pheochromocytoma (control group).

DETAILED DESCRIPTION:
Each patient included in this study underwent unilateral adrenalectomy for adrenal pathology during the inclusion period. For each patient included, intraoperative hemodynamic data were collected every 20 seconds by the monitoring system used by the anesthesia team (VitalSignsCapture v1.004 program via RS232 port). For each patient, the HI score (a clinical tool validated in two previously published articles) was calculated for the intraoperative period (time between induction of anesthesia and patient discharge from the operating room). This enabled a comparison to be made between patients operated on for pheochromocytoma (30 patients) and patients operated on for a cause other than pheochromocytoma (30 patients).

ELIGIBILITY:
Inclusion Criteria:

* Patients operated on for unilateral adrenal pathology by laparosocopic approach (pheochromocytoma and non-pheochromocytoma)

Exclusion Criteria:

* Patients operated on for unilateral adrenal pathology by laparosocopic approach (pheochromocytoma and non-pheochromocytoma)
* Patients operated on for bilateral adrenal pathology

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated on for unilateral adrenal pathology by laparosocopic approach (pheochromocytoma and non-pheochromocytoma) in the department of gastrointestinal, metabolic and cancer surgery (CVMC, CHU Nancy)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Hemodynamic instability score | during surgery (from induction of the patient under general anesthesia to discharge from the operating room)
  The haemodynamic instability score was calculated as a weighted continuous measure ranging from 0 to 160 points. This score appropriately quantifies deviations of blood pressure and heart rate from predefined thresholds, and infusion rates of vasoactive agents and fluids. Zero corresponds to the absence of peroperative hemodynamic changes and 160 to the maximum possible peroperative hemodynamic changes.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brunaud, Principal Investigator — CHU Nancy, Department CVMC
Locations (1):
- CHRU Nancy - Département Chirurgie Viscérale, Métabolique et Cancérologique CVMC (7ème étage), Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Buitenwerf E, Boekel MF, van der Velde MI, Voogd MF, Kerstens MN, Wietasch GJKG, Scheeren TWL. The haemodynamic instability score: Development and internal validation of a new rating method of intra-operative haemodynamic instability. Eur J Anaesthesiol. 2019 Apr;36(4):290-296. doi: 10.1097/EJA.0000000000000941. PMID 30624247
- [Result] Buitenwerf E, Osinga TE, Timmers HJLM, Lenders JWM, Feelders RA, Eekhoff EMW, Haak HR, Corssmit EPM, Bisschop PHLT, Valk GD, Veldman RG, Dullaart RPF, Links TP, Voogd MF, Wietasch GJKG, Kerstens MN. Efficacy of alpha-Blockers on Hemodynamic Control during Pheochromocytoma Resection: A Randomized Controlled Trial. J Clin Endocrinol Metab. 2020 Jul 1;105(7):2381-91. doi: 10.1210/clinem/dgz188. PMID 31714582